CLINICAL TRIAL: NCT04497636
Title: Mental Health Impact of the COVID-19 Pandemic Among Immigrants in Santiago, Chile (STRING-COVID)
Brief Title: Mental Health Impact of the COVID-19 Pandemic Among Migrants in Chile
Acronym: STRING-COVID
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Other Study IDs: 170519004
Record Dates: First submitted 2020-08-01; First posted 2020-08-04 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2020-08

CONDITIONS: Anxiety; Depression; Stress, Psychological; Loneliness; Social Isolation
Keywords: Migrants; Depression; Anxiety; COVID-19; Within-group longitudinal design
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological; Social Isolation; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The mental health of a representative sample of immigrants residing in Santiago, Chile (STRING cohort) was assessed nine months prior to the COVID-19 pandemic (T0). Evidence suggests that social isolation affects mental health by increasing symptoms of anxiety and depression. One of the main components of the current COVID-19 pandemic is the social isolation imposed on the population. This study seeks to explore the short (T1) and long-term (T2) effects of the pandemic on the psychological wellbeing of the cohort.

Specific aims are to

1. Describe the variations in the levels of mental health problems (i.e. symptoms of depression, anxiety, post-traumatic stress, sleep difficulties) and wellbeing of immigrants during the first (T1) and second follow-up (T2)
2. Calculate the short (T1) and long-term (T2) effects of social isolation on the levels of mental health problems of the immigrant population, and
3. Identify risk / protective factors associated with a short (T1) and long-term (T2) increase in mental health problems

DETAILED DESCRIPTION:
Participants were interviewed at baseline (T0) 8 months before the COVID-19 pandemic. An online survey will be applied in two follow-up moments during the pandemic:

1. At 9 months (also 1 month after lockdown measures imposed) (T1)
2. At 18 months (also 10 months after lockdown measures imposed) (T2)

ELIGIBILITY:
Inclusion Criteria:

* Country of birth other than Chile
* Time since arrival to Chile: 3 months (at baseline)

Exclusion Criteria:

* Unable to understand Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The STRING cohort is comonsed of 1,092 adults residing in private households in the Metropolitan Region of Santiago, Chile who were born outside of Chile and had lived in the country for at least 3 months in the first wave.
Sampling Method: Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Month 1 (T1) and month 10 (T2)
  The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) is used to measure symptoms of depression in accordance with the diagnostic criteria for major depressive disorder. The questionnaire consists of nine items scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27. Higher scores indicate greater depression severity, and scores above 10 are considered as the cut-off that indicate that the patient is within the depressive area. Specific cut-off for primary care samples in Chile have been found yielding a cut-off of 7 and above for high sensitivity and specificity (Saldivia, Aslan, Cova, Vicente, Inostroza & Rincón, 2019).
  Changes in depressive symptoms between baseline (T0) and two follow-up points (T1 and T2) will be assessed.
Symptoms of anxiety | Month 1 (T1) and month 10 (T2)
  The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is used to measure symptoms of anxiety and worry. The questionnaire consists of seven items scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21. Specific cut-off for primary care samples in Spain have been found yielding a cut-off of 10 and above for high sensitivity and specificity (García-Campayo et al, 2010).
  Changes in symptoms of anxiety between baseline (T0) and two follow-up points (T1 and T2) will be assessed.

SECONDARY OUTCOMES:
Symptoms of post-traumatic stress disorder | Month 1 (T1) and month 10 (T2)
  The Impact of Events Scale (IES-R; Weiss & Marmar, 1997) is used to measure symptoms of post-traumatic stress disorder (PTSD). There scale consists of 22 questions which are scored on a five-point Likert scale (0=not at all, 1=a little bit, 2=moderately, 3=quite a bit, 4=extremely). There are three subscales (i.e., avoidance, intrusion, hyperarousal) and the sum of the three subscales scores comprise the total score. A total score ≥33 indicates the likely presence of PTSD using criteria from the Diagnostic Symptom Manual (DSM-IV).
  Changes in symptoms of post-traumatic stress between the two follow-up points (T1 and T2) will be assessed.
Changes in sleep difficulties | Month 1 (T1) and month 10 (T2)
  The Insomnia Severity Index (ISI; Bastein CH, et al. 2001) is used to assess the nature, severity, and impact of sleep difficulties. The questionnaire consists of 7 items scored on a five-point Likert scale (0=no problem, 4=very severe problem) with scores ranging from 0 to 28.
  Changes in symptoms sleep difficulties between the two follow-up points (T1 and T2) will be assessed.
Changes in hazardous and harmful alcohol drinking | Month 1 (T1) and month 10 (T2)
  Using the three-item Alcohol Use Disorders Identification Test (AUDIT-C). Changes in hazardous and harmful alcohol drinking between baseline (T0) and two follow-up points (T1 and T2) will be assessed.
Changes in loneliness | Month 1 (T1) and month 10 (T2)
  Using the three-item Revised UCLA Loneliness Scale. Scores range from 3 to 9 with higher scores indicating higher perceived loneliness.
  Changes in perceived loneliness between the two follow-up points (T1 and T2) will be assessed.
Change in general physical and mental health | Change from last 2 weeks before pandemic to month 1 (T1) and month 10 (T2)
  Change in general physical and mental health, self-rated, on a VAS scale from 0 to 100. Higher scores indicate worse self-reported health.
  Changes in perceived general physical and mental health between the two follow-up points (T1 and T2) will be assessed.
Change in mental health symptoms from last 2 weeks before the pandemic to the last 2 weeks during the COVID-19 pandemic at T1 and T2. | Change from last 2 weeks before pandemic to month 1 (T1) and to month 10 (T2).
  Change in visual analogue scale-assessed transdiagnostic measures across all psychiatric symptoms in the last 2 weeks compared to the last 2 weeks of "regular life" before the COVID-19 outbreak.
Change in mental health well-being from last 2 weeks before the pandemic to the last 2 weeks during the COVID-19 pandemic at T1 and T2. | Change from last 2 weeks before pandemic to month 1 (T1) and to month 10 (T2).
  Change in World Health Organization (WHO)-5 well-being in the last 2 weeks compared to the last 2 weeks of "regular life" before the COVID-19 outbreak.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Errazuriz, PhD, Principal Investigator — Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, RM, Chile